CLINICAL TRIAL: NCT02918708
Title: Assessment of Antibody Responses in UK Infants Given Two Doses of 10 or 13 Valent Pneumococcal Conjugate Vaccine (PCV) in Infancy and PCV13 in the Second Year of Life (Study Code: Pneumococcal in New Combinations (PINC))
Brief Title: Assessment of Novel Pneumococcal Conjugate Vaccination Scheduled in UK Infants
Acronym: PINC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding channel amended by UK department of health
Sponsor: Public Health England (Other Government)
Collaborators: Imperial College London (Other); Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PINC trial
Record Dates: First submitted 2016-09-12; First posted 2016-09-29 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2017-01

CONDITIONS: Vaccination; Immunization
Keywords: vaccination; immunisation; pneumococcal; conjugate
MeSH Terms: interventions — PHiD-CV vaccine; 10-valent pneumococcal conjugate vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 2 (Synflorix then Prevenar13) (Active Comparator): PCV10 given at 2 and 4 months of age, PCV13 given at 12 months of age
  Interventions: Biological: Synflorix; Biological: Prevenar13
- group 1 (Prevenar13 only) (Active Comparator): PCV13 given at 2,4 and 13 months of age
  Interventions: Biological: Prevenar13

INTERVENTIONS:
Biological: Synflorix — 10-valent pneumococcal conjugate vaccine
  Other Names: PCV10
  Arms: group 2 (Synflorix then Prevenar13)
Biological: Prevenar13 — 13-valent pneumococcal conjugate vaccine
  Other Names: PCV13

SUMMARY:
The National Vaccine Evaluation Consortium conducts Department of Health funded trials trials to provide information to underpin changes to the national immunisation and vaccination schedule.

This study will assess how different schedules of pneumococcal conjugate vaccines work in providing protection to young infants. It is well established that vaccines can behave differently depending on which order they are given and alongside which other immunisations. This has been shown for Hib and MenC vaccines, which are similar in structure to the pneumococcal vaccines that will be studied here. The investigators will measure responses to the pneumococcal vaccines as well as to other routine immunisations, all of which will be provided by our study team. Infants will be recruited by dedicated study staff through primary care and will participate from their first vaccinations at 2 months of age, until the blood sample taken a month after their boosters at a year old, i.e. until 13 months of age.

Any child found to have antibody levels below that which indicates protection for Hib, MenC, MenB or pneumococcal in the blood sample taken at 13 months of age will be offered an extra dose of the relevant vaccine(s).

DETAILED DESCRIPTION:
The UK Department of Health provides a routine vaccination schedule for children in the UK which is administered by GP surgeries. The schedule is updated by the addition of antigens and amendment of products and schedules over time to improve the protection afforded to the paediatric population and the overall cost-effectiveness of the programme.

It is now well established that the effects of giving different vaccines and antigens together, as well as the order and numbers of doses given for priming and boosting, can affect the immunological responses they elicit. For example co-administration of different polysaccharide conjugate vaccines may enhance responses as shown in a prior study by our group - the National Vaccine Evaluation Consortium (NVEC). This demonstrated that the tetanus-toxoid conjugated MCC vaccine enhanced the response to a co-administered Hib conjugate vaccine if it was also conjugated to tetanus toxoid . In some cases, more than one conjugate vaccine is available for the same disease, as occurred in the early days of the Hib programme when vaccines conjugated to tetanus toxoid or CRM - a natural nontoxigenic diphtheria protein- were both available. NVEC therefore conducted a study to assess the impact of interchanging the two different Hib conjugate vaccines for the three dose primary immunisation course. This showed that interchanging the two different Hib conjugates for primary immunisation did not compromise immune responses and some mixed schedules gave higher antibody responses than those in which all three doses were given with the same conjugate. However, when mixed schedules of MCC-TT and MCC-CRM were subsequently studied by NVEC a MCC-CRM/MCC-TT two dose schedule was shown to be inferior to those in which MCC-TT was given as the first priming dose.

Until now, the UK has used pneumococcal conjugate vaccines from Pfizer in the form of seven or 13 valent PCV, with the current schedule recommending vaccination with PCV13 at 2, 4 and 12 months of age (2+1 schedule). The 13 polysaccharide serotypes in PCV13 are conjugated to CRM. More recently a 10 valent conjugate vaccine manufactured by GSK (PCV10) has been licensed for use in the UK as a 2+1 schedule. The 10 serotypes in PCV10 are also in PCV13 but it lacks serotypes 3, 6A and 19A. No significant protection in vaccinated infants has been shown by PCV13 against serotype 3 [Andrews et al 2014] and for 6A and 19A PCV10 has been shown to provide some cross protection against these serotypes. Like PCV13, PCV10 is safe and efficacious and is in global use. Unlike PCV13, however, the proteins used for conjugation in PCV10 are a mixture of Haemophilus influenzae protein D, tetanus toxoid and diphtheria toxoid. As with Hib and MCC conjugate vaccines, having two PCV products that could be used in the UK schedule would provide reassurance about vaccine supply and could improve cost effectiveness by reducing vaccine cost. However, if PCV10 vaccine is to be considered for use in the UK, particularly if a combination of PCV10 and PCV13 is used in the national schedule, this would require evidence of the adequate immunogenicity of a mixed schedule and this cannot be inferred from the experience with Hib and MCC conjugates.

The results of a clinical trial in which PCV13 was used for the two priming doses at 2 and 4 months followed by a PCV10 booster dose at 12 months has recently been reported. This showed that a protective antibody response post-booster (serotype specific antibody level by ELISA ≥0.35ug/mL) to 9 of the 13 PCV31 serotypes was achieved by at least 97% of infants boosted with PCV10 whereas PCV13 boosted infants achieved at least 97% protective responses to 11 of the 13 serotypes. For 10 of the 13 serotypes the geometric mean concentrations of antibodies were significantly higher in PCV13 boosted infants and for 3 serotypes were higher in PCV10 boosted infants. This study suggests that mixed PCV schedules in which the CRM-based vaccine is given first may not be optimal.

This study will build on this work, and will assess the alternative combination, which will be PCV10 for priming followed by PCV13 for boosting. The comparator arm will be the current standard of care. The study will therefore include two groups:

2+1 : PCV13 at 2, 4 and 12 months of age 2+1 PCV10 at 2 and 4 months of age followed by PCV13 at 12 months of age

All participants will receive all other vaccines as defined under the routine infant immunisation schedule.

This study will rapidly provide information to the JCVI on options for the UK schedule for pneumococcal immunisation of infants and how best the current options could be expanded whilst retaining appropriate protection as afforded through the current schedule.

This study is funded by the UK Department of Health and sponsored by Public Health England. Following written informed consent from their parent/ guardian, infants will be randomly assigned to one of the two treatment groups and will receive all their vaccinations to 12 months of age as well as having two blood samples. The first sample will be a month after completion of the primary series, at about five months of age, and the second a month after the booster doses, at about 13 months of age. Extra doses of MenB, MenC, Hib and/or pneumococcal vaccine(s) will be offered where the immune response measured in the post-booster blood is below the correlate of protection.

Information from the study will be presented to the Department of Health to underpin ongoing evolution of the national vaccination schedule. A manuscript will be submitted for publication to a peer reviewed journal and all participating families will receive a summary of the study findings by post.

ELIGIBILITY:
Inclusion Criteria:

* Infants due to receive their primary immunisations , aged up to 13 weeks on first vaccinations.
* Written informed consent given by mother who is aged ≥>= 16 years [NB mother is preferable as consent also allows permission to record the date of pertussis immunisation in pregnancy, which may need to be verified in her medical record. Where mother is not available, consent may be taken from father or legal guardian and maternal pertussis status noted as not known]

Exclusion Criteria:

* Bleeding disorder
* Fulfil any of the contraindications to vaccination as specified in The Green Book [https://www.gov.uk/government/organisations/public-health-england/series/immunisation-against-infectious-disease-the-green-book]

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
pneumococcal proportions | 13 months of age
  proportions with protective antibody levels to each serotype in the pneumococcal conjugate vaccine

SECONDARY OUTCOMES:
pneumococcal GMC | 13 months of age
  geometric mean concentration of each serotype included in pneumococcal conjugate vaccine
pneumococcal fold rise | 13 months of age
  to estimate fold rises in antibody for each serotype included in pneumococcal conjugate vaccine
Men B proportions | 5 and 13 months of age
  to estimate proportions with protective antibody levels against the three strains included in the vaccine
Men B GMT | 5 and 13 months of age
  to estimate the geometric mean titres of serum bactericidal antibody levels
tetanus proportions | 5 months of age
  to estimate proportions achieving the protective antibody levels
tetanus GMC | 5 months of age
  to estimate the geometric mean concentration of antibody levels against tetanus
diphtheria GMC | 5 months of age
  to estimate the geometric mean concentration of antibody levels against diphtheria
diphtheria proportions | 5 months of age
  to estimate proportions achieving the protective antibody levels
pertussis GMC | 5 months of age
  to estimate the geometric mean titres of antibody levels against pertussis components
MenC proportions | 13 months of age
  to estimate proportions achieving the protective antibody levels
MenC GMT | 13 months of age
  to estimate the geometric mean titres of antibody levels against MenC
Hib proportions | 5 and 13 months of age
  to estimate proportions achieving the protective antibody levels
Hib GMC | 5 and 13 months of age
  to estimate the geometric mean concentration of antibody levels against Hib
reactogenicity | one week after each vaccination
  Assessment of reactogenicity of vaccines from parent completed health diaries for the week following each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Chair — Public Health England
Locations (2):
- United Kingdom (2):
  - Hertfordshire primary care, Hertfordshire, Hertfordshire
  - Imperial Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No